CLINICAL TRIAL: NCT03702985
Title: A Phase II Trial of Capecitabine and Irinotecan With or Without Amifostine in Neoadjuvant Chemoradiotherapy in Locally Advanced Rectal Cancer
Brief Title: Radiation-protection Effect of Amifostine in Locally Advanced Rectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhu Ji, professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FDRT-R007
Record Dates: First submitted 2018-06-14; First posted 2018-10-11 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2018-10

CONDITIONS: Locally Advanced Rectal Cancer
Keywords: Neoadjuvant Chemoradiotherapy; amifostine; irinotecan; capecitabine
MeSH Terms: interventions — Radiation; Capecitabine; Irinotecan; Amifostine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Capecitabine and Irinotecan without Amifostine (Active Comparator): Concurrent Chemoradiotherapy:
  Radiation: 50Gy/25Fx; Capecitabine: 625mg/m2 bid Monday-Friday per week; Irinotecan: 80mg/m2 (UGT1A1*28 6/6) or 65mg/m2 (UGT1A1*28 6/7)
  Chemotherapy in Interval Between CRT and Surgery:
  Capecitabine: 1000mg/m2 bid d1-14; Irinotecan: 200mg/m2 d1
  Surgery:
  Scheduled 6-8 weeks after the completion of CRT Adjuvant Chemotherapy: depends on patients pathological review.
  Interventions: Radiation: Radiation; Drug: Capecitabine; Drug: Irinotecan
- Capecitabine and Irinotecan with Amifostine (Experimental): Concurrent Chemoradiotherapy:
  Radiation: 50Gy/25Fx; Capecitabine: 625mg/m2 bid Monday-Friday per week; Irinotecan: 80mg/m2 (UGT1A1*28 6/6) or 65mg/m2 (UGT1A1*28 6/7) Amifostine: 400mg/m2 per week
  Chemotherapy in Interval Between CRT and Surgery:
  Capecitabine: 1000mg/m2 bid d1-14; Irinotecan: 200mg/m2 d1
  Surgery:
  Scheduled 6-8 weeks after the completion of CRT Adjuvant Chemotherapy: depends on patients pathological review.
  Interventions: Radiation: Radiation; Drug: Capecitabine; Drug: Irinotecan; Drug: Amifostine

INTERVENTIONS:
Radiation: Radiation — Pelvic Radiation: 50Gy/25Fx
Drug: Capecitabine — 625mg/m2 bid Monday-Friday per week
  Other Names: Xeloda
Drug: Irinotecan — 80mg/m2 (UGT1A1*28 6/6) or 65mg/m2 (UGT1A1*28 6/7)
Drug: Amifostine — 400mg/m2 per week
  Arms: Capecitabine and Irinotecan with Amifostine

SUMMARY:
The study evaluates the addition of Amifostine to capecitabine and irinotecan in neoadjuvant chemoradiation(CRT) in locally advanced rectal cancer. Half of participants will receive capecitabine and along with neoadjuvant radiotherapy, followed by a cycle of XELIRI, while the others will receive capecitabine and irinotecan added by amifostine during CRT, followed by a cycle of XELIRI. All participants will be scheduled to receive surgery 6-8 weeks after the completion of CRT. Then it will depends which regimens the patient would receive according to his or her pathological results.

ELIGIBILITY:
Inclusion Criteria:

* pathological confirmed adenocarcinoma
* clinical stage T3-4 and/or N+
* the distance from anal verge less than 12 cm
* without distance metastases
* performance status score: 0~1
* UGT1A1*28 6/6 or 6/7
* without previous anti-cancer therapy
* sign the inform consent

Exclusion Criteria:

* pregnancy or breast-feeding women
* serious medical illness
* baseline blood and biochemical indicators do not meet the following criteria: neutrophils≥1.5×10^9/L, Hb≥90g/L, PLT≥100×10^9/L, ALT/AST ≤2.5 ULN, Cr≤ 1 ULN
* DPD deficiency
* UGT1A1*28 7/7

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2018-05-28 (Actual); Primary Completion 2019-11-01 (Estimated); Study Completion 2020-03-01 (Estimated)

PRIMARY OUTCOMES:
the morbidity of hematological adverse events and diarrhea as assessed by CTCAE v4.0 | during neoadjuvant chemoradiation.

SECONDARY OUTCOMES:
Impact of participants' quality of life during treatment as assessed by EQ-5D questionnaire and EORTC-QLQ-C30 questionnaire | during neoadjuvant chemoradiation.
pathological response rate | Surgery scheduled 6-8 weeks after the end of chemoradiation.
the morbidity of late radiation proctitis | late radiation proctitis is measured 9 months after the end of chemoradiation.

CONTACTS AND LOCATIONS:
Overall Officials: Zhen Zhang, MD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China